CLINICAL TRIAL: NCT06590467
Title: Abbott Structural Heart Device Registry
Acronym: SH-Registry
Status: Recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10415
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-01

CONDITIONS: Heart Diseases; ASD - Atrial Septal Defect; VSD - Muscular Ventricular Septal Defect; PFO - Patent Foramen Ovale; PIVSD - Post Infarct Muscular Ventricular Septal Defect; Valvular Heart Disease
Keywords: Amplatzer; Amplatzer Septal Occluder; Amplatzer Multi-fenestrated (Cribriform) Occluder; Amplatzer Duct Occluder; Amplatzer Piccolo Occluder; Amplatzer Muscular VSD Occluder; Amplatzer Post-Infarct VSD Occluder; Amplatzer Talisman; Amplatzer TorqVue Delivery System; Amplatzer Sizing Balloon; Amplatzer Guidewire; Amplatzer Occluder devices; Surgical Valves; Epic Plus Aortic Valve; Epic Plus Mitral Valve; Epic Plus Supra Aortic Valve; Epic Max Aortic Valve; Bioprosthetic heart valve; Surgical tissue heart valve
MeSH Terms: conditions — Heart Diseases; Heart Septal Defects, Atrial; Foramen Ovale, Patent; Heart Valve Diseases | interventions — Septal Occluder Device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Amplatzer: * ASO: ≥50 cases/year
  * ASD-MF: ≥50 cases/year
  * ADO: ≥50 cases/year
  * ADO II: ≥50 cases/year
  * Piccolo: ≥50 cases/year
  * MuVSD: Up to 50 cases/year
  * PI-VSD: Up to 50 cases/year
  * Talisman/TDS: ≥100 cases/year
  * TorqVue Delivery Systems Group 1 (ATV/ITV/EITV/TV2): 250 cases/year across different occluders
  * TorqVue Delivery Systems Group 2 (TVLP/TVLPC): 100 cases/year across different occluders
  * SB II:100 PFO cases/year & 100 ASD cases/year
  * GW: 200 cases/year
  Interventions: Device: Amplatzer™ Occlusion Devices
- Cardiac Surgery: It is anticipated that approximately 830 subjects implanted with at least one applicable Abbott surgical tissue heart valve (THV) will be enrolled and followed for 10 years.
  * Approximately 225 subjects receiving Epic Plus mitral valves
  * Approximately 150 subjects receiving Epic Plus aortic valves
  * Approximately 170 subjects receiving Epic Plus Supra aortic valves
  * Approximately 285 subjects receiving Epic Max aortic valves
  Interventions: Device: Epic™ Surgical Tissue Heart Valve devices

INTERVENTIONS:
Device: Amplatzer™ Occlusion Devices — The Amplatzer™ Occluders are devices intended for the occlusion of multiple septal heart defects.
  Other Names: Amplatzer Septal Occluder; Amplatzer Multi-fenestrated (Cribriform) Occluder; Amplatzer Duct Occluder; Amplatzer Piccolo Occluder; Amplatzer Muscular VSD Occluder; Amplatzer Post-Infarct VSD Occluder; Amplatzer Talisman; Amplatzer TorqVue Delivery System
  Groups: Amplatzer
Device: Epic™ Surgical Tissue Heart Valve devices — The Epic™ valves are indicated for patients requiring replacement of a diseased, damaged, or malfunctioning native aortic/mitral heart valve. It may also be used as a replacement for a previously implanted aortic/mitral prosthetic heart valve.
  Other Names: EMAX; E200; ESP200; Sizer Set Model E2000; Sizer Set Model EMAX-1000; Replacement Holder Handles E2000-HA and E2000-HM
  Groups: Cardiac Surgery

SUMMARY:
The Abbott Structural Heart (SH) Registry is being conducted to confirm the safety and performance of Abbott's SH devices in a post-market, real-world setting. The Registry primarily involves gathering data from routine hospital practices and standard-of-care (SOC) procedures administered to patients. All devices used in these procedures must be commercially available to the participating site. A list of specific devices covered by the Registry are available upon request from the Sponsor. Data generated by the Registry will be used to meet regulatory requirements, such as the European Union Medical Device Regulations 2017/745, that require active post-market clinical follow-up (PMCF) for all commercially available devices.

DETAILED DESCRIPTION:
The Abbott SH Device Registry is designed to confirm the safety and performance of commercially available Abbott SH devices as they are used in routine hospital practice or SOC procedures. Patients will be screened for eligibility and willingness to participate prior to the procedure or, if enrolled retrospectively, within the following timeframes:

* Amplatzer portion: within 7 days post-procedure
* Cardiac Surgery portion: within 6 months post-procedure.

All patients who provide informed consent and undergo an implant attempt with an applicable Abbott SH device are eligible to participate in the Registry. The Registry anticipates that approximately 500 subjects per year will be enrolled. The projected enrollment period is at least 5 years.

The Registry will be conducted at approximately 25 sites worldwide. Additional sites may be approached for participation in the Registry as needed.

Follow-up visits should align with the site's routine SOC visits for the associated procedure. Data collection will occur post-screening and consent and at post-procedure SOC follow-up visit(s). Where applicable, follow-up visits may occur over the telephone, virtually, or in-office, following SOC practice.

The follow-up duration will depend on the Abbott device(s) used during the procedure. Certain devices will utilize data collection at discharge (or 7 days post procedure, whichever comes first), short-term (1 - 3 months as applicable), a mid-term (6 months), and long-term follow-up (12 months) visits to support clinical safety and performance data requirements. Alternatively, some devices will have follow-up visits extending up to 10 years to monitor subjects throughout the devices' lifetime.

A surgical valve-specific "Line Extension Sub-Study" is included in the protocol to collect data at European sites with the intention of applying for approval in the US for 2 specific surgical aortic valve sizes (Epic Max 27mm, and the Epic Plus Supra 29mm).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is expected to undergo an implant attempt using one or more Abbott Structural Heart devices covered in this Registry or has previously undergone an implant attempt within the timeframes specified in the device-specific appendices.
2. Subject is willing and able to comply with the site's standard of care follow-up schedule.
3. Subject is willing to provide appropriate informed consent for Registry participation. For deceased subjects enrolled retrospectively, local regulations and EC/IRB recommendations regarding consent and the protection of personal data must be followed.

Exclusion Criteria:

1. Subject is participating in another clinical study that would affect the results of this Registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This Registry is open to enroll subjects of all genders and ages from the general population who undergo a procedure that use at least one Abbott SH device included in this Registry (including unsuccessful implants). Subjects must meet all eligibility criteria and provide written informed consent prior to sites conducting any investigation-specific procedures not considered standard of care.
  Patients will be screened for eligibility and willingness to participate prior to the procedure or, if enrolled retrospectively, within the timeframe specified in the device-specific appendices of the protocol (Amplatzer cohort: consent within 7days of procedure // Cardiac Surgery cohort: consent within 6 months (183 days) of the implant procedure)
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2039-11 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 7 days
  The primary safety endpoint will be the proportion of subjects with device- and/or procedure-related serious adverse events (SAEs) occurring within 7 days of the procedure.
Primary Effectiveness Endpoint | Baseline
  The primary effectiveness endpoint will be the proportion of procedures that achieved technical success, defined as completion of the procedure with an applicable Abbott SH device implanted

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Abbott
Locations (27):
- United States (4):
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Mount Sinai Hospital, New York, New York
  - UPMC, Pittsburgh, Pennsylvania
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Odense University Hospital, Odense, Southern Denmark, Denmark
- Tartu University Hospital, Tartu, Tartu, Estonia
- France (3):
  - CHRU Hopital de Pontchaillou, Rennes, Brittan
  - Centre Médico Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Hopital Haut Leveque, Pessac
- Germany (6):
  - Deutsches Herzzentrum München des Freistaates Bayern, München, Bavaria
  - Klinikum Links der Weser, Bremen, City state Bremen
  - Universitatsklinikum Jena, Jena, Germany
  - Städt. Klinikum Braunschweig gGmbH, Braunschweig, L Saxon
  - Deutsches Herzzentrum der Charité, Berlin, State of Berlin
  - Schüchtermann-Schiller´sche Kliniken GmbH & Co. KG, Bad Rothenfelde
- Children's Health Ireland (CHI), Crumlin, Dublin, Ireland
- Italy (4):
  - IRCCS Policlinico San Donato - Cardio, San Donato Milanese, Lombardy
  - Policlinico San Donato, San Donato Milanese, Lombardy
  - A.O.U. Citta della Salute e della Scienza di Torino, Turin, Piedmont
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- Slaskie Centrum Chorob Serca, Zabrze, Silesian Voivodeship, Poland
- Spain (4):
  - Hospital Infantil Sant Joan De Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Virgen de Rocio, Seville, Spain
  - Hospital Universitario de la Paz - Pediatrico, Madrid
- United Kingdom (2):
  - Royal Brompton Hospital, London, UK
  - St. Thomas Hospital, London